CLINICAL TRIAL: NCT04152408
Title: A Study to Investigate the Function, Safety and Tolerability of the FiberSense System in Diabetic Patients for a Period of Continuous Blood Glucose Monitoring up to 30 Days
Brief Title: Clinical and Home Use Feasibility Study of a Percutaneous Optical Glucose Fiber Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeSense GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P-4.3-C-01
Record Dates: First submitted 2018-10-22; First posted 2019-11-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetes (DM)
Keywords: diabetes management; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FiberSense System (Experimental): 6 diabetic patients will wear a FiberSense system at the upper arm for up to 30 days. and a comparator CGM system at the abdomen (replaced every 7 days).
  Interventions: Device: FiberSense System

INTERVENTIONS:
Device: FiberSense System — FiberSense system, a novel CGM system, based on a fiber-optical sensor placed through the dermis of the patient.

SUMMARY:
This is a single-centre, open label (unblinded) prospective study investigating the performance and safety of FiberSense system in diabetic patients (Typ I and II). In the period of up to 30 days the performance of the FiberSense system is evaluated against laboratory gold standard method during 6 in-clinic sessions.

DETAILED DESCRIPTION:
The FiberSense system is intended to be used by diabetic patients in a home use setting as a CGM system using the interstitial fluid (ISF) glucose as an indicator of blood glucose levels.The purpose of this study is to assess the performance of FiberSense system across the glucose measurement ranges as compared with a laboratory standard reference method in diabetic patients (Type I and II) during in-clinic glucose challenge sessions. At the same time the blood glucose values are recorded by comparator continuous glucose monitoring (CGM) system and self-monitoring blood glucose system (SMBG). The safety aspects are also investigated during the wearing time of up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years old.
* Type I or II diabetes mellitus.
* Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study. If of child bearing potential, the patient must agree to abstain from sexual intercourse or use reliable forms of contraception (e.g. condom or diaphragm with spermicide or oral contraceptives) to prevent pregnancy for the length of the clinical study.
* Willingness, ability and commitment to comply with the testing procedure and follow-up outlined in this protocol including (but not limited to) frequency of clinic visits, use of pre-specified glucose monitoring device.
* Willingness to abstain from swimming during their participation in the measurement phase.
* Willingness to abstain from air travelling during their participation in the measurement phase.
* Willingness to avoid strong magnetic and electrical fields as well as proximity to sensitive medical devices due to the possible electromagnetic interference during their participation in the measurement phase.
* In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a good study candidate.
* Written informed consent to participate in the study provided by the patient.

Exclusion Criteria:

* Poorly controlled diabetes mellitus with HbA1C >10%.
* Known microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as e.g. history of laser coagulation, proliferative diabetic retinopathy, known diabetic nephropathy (with glomerular filtration rate (eGFR) < 45 ml/min) or neuropathy requiring treatment.
* History of significant hypoglycemia unawareness, or a history of severe hypoglycemia (requiring emergency medical intervention) within the last 6 months.
* Currently pregnant, as demonstrated by a positive pregnancy test at screening and prior to enrollment.
* Impaired hepatic function measured as aspartate aminotransferase (AST) ≥ three times the upper reference limit.
* Impaired renal function measured as creatinine > 1.2 times above the upper limit of normal.
* Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
* Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
* Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
* Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
* Have a known allergy to medical-grade adhesives, or known hypersensitivity to any of the products used in the study.
* Known current or recent alcohol or drug abuse
* Blood donation of more than 500 ml within the last three months
* Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
* Has a MRI scan, CT scan, diathermy or flight scheduled during the proposed study participation.
* An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Performance of the FiberSense system as compared with laboratory gold standard reference (LGSR) | at 1, 3, 7, 14, 21 and 28 days
  Point accuracy of the FiberSense system as determined by proportion of CGM readings within ≤15% of the LGSR reading for blood glucose levels >100 mg/dl, and within ≤15 mg/dl of the LGSR reading for blood glucose levels ≤100 mg/dl, for paired samples taken during the in-clinic sessions.
Duration of use of the FiberSense system | 30 days
  Duration of use of the FiberSense device in average and by individual patients
Incidence of (Serious) Adverse Events | 30 days
  Adverse Events reporting and local tolerability as assessed by Draize's scale

SECONDARY OUTCOMES:
Mean and Median Relative Differences in FiberSense measured glucose from LGSR | at 1, 3, 7, 14, 21 and 28 days
Mean and Median Absolute Relative Differences in FiberSense measured glucose from reference laboratory standard | at 1, 3, 7, 14, 21 and 28 days
Hypoglycemia (<75 mg/dl (14)) and hyperglycemia (>180 mg/dl (14)) detection rates | at 1, 3, 7, 14, 21 and 28 days
Hypoglycemia (<75 mg/dl) and hyperglycemia (>180 mg/dl,) missed detection rates | at 1, 3, 7, 14, 21 and 28 days
Accuracy of glucose rate of change of FiberSense sensor compared to glucose rate of change of reference laboratory standard | at 1, 3, 7, 14, 21 and 28 days
Lag time between FiberSense readings and reference laboratory standard results during induced glucose excursions | at 1, 3, 7, 14, 21 and 28 days
Agreement and accuracy relative to SMBG readings (same model to be used by all patients) | weekly - Days 7, 14, 21, 28
  Performance of SMBG evaluated as percentage of system readings within 15%, 20%, 30% and 40% of LGSR values and by means of MARD and MedARD(%)
Stability of the FiberSense fluorescence measurements | weekly - Days 7, 14, 21, 28
  The stability of sensor performance over the 30-day time period evaluated as percentage of FiberSense system readings within 15%, 20%, 30% and 40% of LGSR values and by means of MARD and MedARD(%)
User satisfaction assessed by the Likert scale | 30 days
  Subjective impression of the patients on the scale of 1 (strongly agree) to 5 (strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hasslacher, Prof. Dr., Principal Investigator — Diabetes Institut Heidelberg, Germany
Locations (1):
- Diabetes Institut Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No